CLINICAL TRIAL: NCT03781479
Title: A Randomized, Placebo-Controlled, Crossover Study to Evaluate the Safety and Efficacy of Amifampridine Phosphate in Ambulatory Patients With Spinal Muscular Atrophy (SMA) Type 3
Brief Title: Controlled Trial to Evaluate Amifampridine Phosphate in Spinal Muscular Atrophy Type 3 Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalyst Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMA-001
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Results first posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Muscular Atrophy, Spinal
Keywords: Type 3
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Amifampridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Amifampridine Phosphate - Placebo (Experimental): Oral tablets, 30 to 80 mg per day in divided doses 3 to 4 times a day for 4 weeks
  Interventions: Drug: Amifampridine Phosphate; Drug: Placebo Oral Tablet
- Placebo - Amifampridine Phosphate (Experimental): Oral tablets, 30 to 80 mg per day in divided doses 3 to 4 times a day for 4 weeks
  Interventions: Drug: Amifampridine Phosphate; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Amifampridine Phosphate — Amifampridine phosphate tablets 10 mg will be provided in round, white-scored tablets, and containing amifampridine phosphate formulated to be the equivalent of 10 mg amifampridine base per tablet.
  Other Names: 3,4 diaminopyridine phosphate
Drug: Placebo Oral Tablet — Placebo Oral Tablet

SUMMARY:
A two-period, two-treatment, crossover study to evaluate the safety, tolerability and efficacy of amifampridine phosphate in ambulatory patients diagnosed with spinal muscular atrophy (SMA) Type 3.

DETAILED DESCRIPTION:
This randomized (1:1), double-blind, placebo-controlled, 2-period, 2-treatment, crossover, outpatient study is designed to evaluate the safety, tolerability and efficacy of amifampridine phosphate in ambulatory patients diagnosed with SMA Type 3. The study is planned to include approximately 12 male and female SMA Type 3 patients. The planned duration of participation for each patient is approximately 2 months, based upon length of dose titration and excluding the screening period, which can last up to 14 days. Patients should only be taking the assigned investigational product (amifampridine phosphate 10 mg tablets or matching placebo tablets), no new therapies are permitted during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent after the nature of the study has been explained and before the start of any research-related procedures.
2. Male or female between the ages of 6 and 50 years.
3. Genetically confirmed diagnosis of SMA Type 3.
4. Able to walk independently for at least 30 meters.
5. Not taking Nusinersen for the treatment of SMA (Nusinersen should be stopped at least 6 months before screening). Salbutamol is permitted only if the dose has been stable during the 6 months before screening.
6. Able to swallow oral medication.
7. Female patients of childbearing potential must have a negative pregnancy test (serum human chorionic gonadotropin [HCG] at Screening); and must practice an effective, reliable contraceptive regimen during the study and for up to 30 days following discontinuation of treatment.
8. Ability to participate in the study based on overall health of the patient and disease prognosis, as applicable, in the opinion of the Investigator; and able to comply with all requirements of the protocol, including completion of study questionnaires.

Exclusion Criteria:

1. Epilepsy and currently on medication for epilepsy.
2. Concomitant use of medicinal products with a known potential to cause QTc prolongation.
3. Patients with long QT syndromes.
4. An electrocardiogram (ECG) within 6 months before starting treatment that shows clinically significant abnormalities, in the opinion of the Investigator.
5. Breastfeeding or pregnant at Screening or planning to become pregnant at any time during the study.
6. Treatment with an investigational drug (other than amifampridine), device, or biological agent within 6 months prior to Screening or while participating in this study.
7. Surgery for scoliosis or joint contractures within the previous 6 months.
8. Any medical condition that, in the opinion of the Investigator, might interfere with the patient's participation in the study, poses an added risk for the patient, or confound the assessment of the patient.
9. History of drug allergy to any pyridine-containing substances or any amifampridine excipient(s).
10. Less than a 3-point improvement in HFSME from start of the Open label Run -in period to end of Run-in (Day 0).

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Maggi, MD, Principal Investigator — Carlo Besta Institute, Milan, Italy
Locations (1):
- Neurological Institute Carlo Besta, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bonanno S, Giossi R, Zanin R, Porcelli V, Iannacone C, Baranello G, Ingenito G, Iyadurai S, Stevic Z, Peric S, Maggi L. Amifampridine safety and efficacy in spinal muscular atrophy ambulatory patients: a randomized, placebo-controlled, crossover phase 2 trial. J Neurol. 2022 Nov;269(11):5858-5867. doi: 10.1007/s00415-022-11231-7. Epub 2022 Jun 28. PMID 35763114

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 14 January 2019 - 17 September 2020 at two sites in Europe.
Pre-assignment Details: A screening visit was conducted to ensure that each patient met inclusion/exclusion criteria for the study. Those patients successfully completing screening had procedures/assessments conducted at the start of the Run-in period (Day 1, before starting study medication) and during Run-in, until stable dose and frequency of amifampridine was established for at least 7 days, and at least a 3-point improvement in HFMSE score was achieved from start of Run-in to be eligible for randomization (Day 0).
Groups:
- Amifampridine Phosphate - Placebo: Each patient participated in an open-label unblinded drug escalation/treatment run-in phase for up to 4 weeks until stable dose and frequency of amifampridine phosphate was achieved for 7 days. After this phase, half of the subjects were randomized to receive amifampridine in Period 1 and then crossed over to receive placebo in Period 2. Each randomized treatment period was 14 days in duration.
  Dosing was up to 80 mg per day and frequency was between 3-4 times per day.
  Amifampridine Phosphate: Amifampridine phosphate tablets 10 mg were provided in round, white-scored tablets, and contained amifampridine phosphate formulated to be the equivalent of 10 mg amifampridine base per tablet.
  Placebo: A placebo equivalent was provided as tablets indistinguishable from the amifampridine phosphate tablets. The placebo was administered consistent with the dose and dose regimen of amifampridine phosphate.
- Placebo - Amifampridine Phosphate: Each patient participated in an open-label unblinded drug escalation/treatment run-in phase for up to 4 weeks until stable dose and frequency of amifampridine phosphate was achieved for 7 days. After this phase, half of the subjects were randomized to receive placebo in Period 1 and then crossed over to receive amifampridine in Period 2. Each randomized treatment period was 14 days in duration.
  Dosing was up to 80 mg per day and frequency was between 3-4 times per day.
  Placebo: A placebo equivalent was provided as tablets indistinguishable from the amifampridine phosphate tablets. The placebo was administered consistent with the dose and dose regimen of amifampridine phosphate.
  Amifampridine Phosphate: Amifampridine phosphate tablets 10 mg were provided in round, white-scored tablets, and contained amifampridine phosphate formulated to be the equivalent of 10 mg amifampridine base per tablet.
- Not Randomized: Patients receiving amifampridine during the open-label run-in period but were not randomized to receive treatment.
Period: Overall Study
Arm/Group | Amifampridine Phosphate - Placebo | Placebo - Amifampridine Phosphate | Not Randomized
Started | 6 | 6 | 1
Completed | 6 | 6 | 0
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis of baseline characteristics included all patients in the Safety population, who are those patients who enrolled and received at least one dose of amifampridine. Patients who began the Run-in period regardless of whether they were randomized to double blind medication on Day 0 belong to the Safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Amifampridine Phosphate - Placebo | Placebo - Amifampridine Phosphate | Not Randomized | Total
Number analyzed (Participants) | 6 | 6 | 1 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (8.5) | 30.2 (13.5) | 45.0 | 34.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 0 | 5
  Male | 2 | 5 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 5 | 1 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 64.7 (9.3) | 67.8 (11.8) | 76.9 | 67.0 (10.2)
Height [Mean (Standard Deviation); unit: cm] | 169.3 (9.0) | 174.8 (6.1) | 170.0 | 171.9 (7.6)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.5 (1.4) | 22.3 (4.3) | 26.6 | 22.7 (3.1)

OUTCOME MEASURES:

1. Primary Outcome: Hammersmith Functional Motor Scale Expanded (HFMSE) Summary Statistics and Mixed Model Analysis
Description: Hammersmith Functional Motor Scale Expanded (HFMSE) assesses motor function by functional item in order of progressive difficulty, with higher values showing higher function abilities. Each item is scored on a scale of 0-2 with 2 representing item achieved unaided and 0 representing inability to achieve item. Each item was assessed by the patient at Screening, the first (Day 1) and last day (Day 0) of the Run-in period, during Period 1 at Day 7 and Day 14, and during Period 2 at Day 21 and Day 28. The total HFMSE score was calculated as the sum of each item score, with a maximum score of 66 (all items achieved unaided) and minimum score of 0 (all items failed). Change from baseline (CFB) will be assessed from Day 0 to Day 28. A mixed effects liner model was fit with the HFMSE change from baseline (CFB) scores at Day 28 as a response and treatment, sequence, and treatment by sequence as fixed effect terms and patient as a random effect.
Time Frame: Screening, the first (Day 1) and last day (Day 0) of the Run-in period, during Period 1 at Day 7 and Day 14, and during Period 2 at Day 21 and Day 28
Population: The analysis of primary outcome data was based on the Full Analysis Set population, which included all randomized patients who received at least one dose of study medication (amifampridine or placebo) and had at least one post-treatment efficacy assessment. Patients are compared for efficacy according to the treatment to which they were randomized, regardless of the treatment actually received.
Measure: Least Squares Mean (Standard Error); unit: Overall Score
Groups:
- Amifampridine Phosphate: Each patient will participate in an open-label unblinded drug escalation/treatment run-in phase for up to 4 weeks until stable dose and frequency of amifampridine phosphate is achieved for 7 days. After this phase, half of the subjects were randomized to receive amifampridine in Period 1 and then crossed over to receive placebo in Period 2 and the other were randomized to receive placebo in Period 1 and then crossed over to receive amifampridine in Period 2.
  Each randomized treatment period is 14 days in duration.
  Dosing was up to 80 mg per day and frequency was between 3-4 times per day.
  Amifampridine Phosphate: Amifampridine phosphate tablets 10 mg were provided in round, white-scored tablets, and contained amifampridine phosphate formulated to be the equivalent of 10 mg amifampridine base per tablet.
  Placebo: A placebo equivalent was provided as tablets indistinguishable from the amifampridine phosphate tablets. The placebo was administered consistent with the dose and dose regimen of amifampridine phosphate.
  The Amifampridine study arm includes all patients in the FAS population who received Amifampridine during the treatment period, regardless of which Period the treatment was administered.
- Placebo: Each patient will participate in an open-label unblinded drug escalation/treatment run-in phase for up to 4 weeks until stable dose and frequency of amifampridine phosphate is achieved for 7 days. After this phase, half of the subjects were randomized to receive amifampridine in Period 1 and then crossed over to receive placebo in Period 2 and the other were randomized to receive placebo in Period 1 and then crossed over to receive amifampridine in Period 2.
  Each randomized treatment period is 14 days in duration.
  Dosing was up to 80 mg per day and frequency was between 3-4 times per day.
  Amifampridine Phosphate: Amifampridine phosphate tablets 10 mg were provided in round, white-scored tablets, and contained amifampridine phosphate formulated to be the equivalent of 10 mg amifampridine base per tablet.
  Placebo: A placebo equivalent was provided as tablets indistinguishable from the amifampridine phosphate tablets. The placebo was administered consistent with the dose and dose regimen of amifampridine phosphate.
  The Placebo study arm includes all patients in the FAS population who received Placebo during the treatment period, regardless of which Period the treatment was administered.
Arm/Group | Amifampridine Phosphate | Placebo
Number analyzed (Participants) | 12 | 12
Overall Score | 0.208 (0.326) | -0.583 (0.326)
Statistical Analysis 1: Comparison: Amifampridine Phosphate vs Placebo; A mixed effects liner model was fit with the HFMSE change from baseline (CFB) scores at Day 28 as a response and treatment, sequence, and treatment by sequence as fixed effect terms and patient as a random effect; Test type: Other; p = 0.0083, Mixed Models Analysis; Mean Difference (Net) = 0.792, 95% CI 2-sided [0.22 to 1.37] — Results show the LSMeans for the estimated difference between treatments along with a 95% confidence interval for this difference

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were recorded for each patient from the time informed consent was obtained at Screening and continued through four weeks after the last visit or at the early discontinuation visit, for a total of approximately 14 weeks. Non-serious AEs were recorded for each patient after the first administration of study drug through the termination visit or at the early termination visit, for a total of approximately 10 weeks.
Description: Serious classification based on the FDA regulatory definition of a serious AE.
Groups:
- Amifampridine; Placebo: Treatment administered to the patient at the time of onset of the AE.
Arm/Group | Amifampridine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amifampridine (N=12) | Placebo (N=12)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 3 | 0
Fatigue (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Transaminases increased (Investigations) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Intranasal Paraesthesia (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT03781479/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT03781479/SAP_001.pdf